CLINICAL TRIAL: NCT04833582
Title: A Phase 1/2 Dose Escalation and Dose Expansion Study of ZN-c3 in Combination With Gemcitabine in Adult and Pediatric Subjects With Relapsed or Refractory Osteosarcoma
Brief Title: A Study of ZN-c3 in Combination With Gemcitabine in Subjects With Osteosarcoma
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: K-Group, Beta, Inc., a wholly owned subsidiary of Zentalis Pharmaceuticals, Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: ZN-c3-003
Record Dates: First submitted 2021-03-25; First posted 2021-04-06 (Actual); Last update posted 2023-11-14 (Actual); Status verified 2023-11

CONDITIONS: Osteosarcoma
MeSH Terms: conditions — Osteosarcoma | interventions — Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Combination ZN-c3 with Gemcitabine (Experimental)
  Interventions: Drug: ZN-c3; Drug: Gemcitabine

INTERVENTIONS:
Drug: ZN-c3 — ZN-c3 is an investigational drug.
Drug: Gemcitabine — Gemcitabine is an approved drug
  Other Names: Gemzar

SUMMARY:
This is a phase 1/2 study of ZN-c3 in combination with gemcitabine in adult and pediatric subjects with relapsed or refractory osteosarcoma.

DETAILED DESCRIPTION:
This is a phase 1/2 dose escalation and dose expansion study, evaluating the clinical activity and safety, pharmacodynamics, and pharmacokinetics of ZN-c3 in combination with gemcitabine in relapsed or refractory osteosarcoma.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 12 years at the time of informed consent
* Bodyweight ≥ 40 kg
* Histologically documented relapsed or metastatic osteosarcoma.
* Must have measurable disease according to RECIST Guideline version 1.1 criteria.
* Adequate hematologic and organ function.
* Female subjects of childbearing potential and male subjects must agree to use an effective method of contraception per institutional standard prior to the first dose and for 6 months after study treatment discontinuation.
* Willingness and ability to comply with scheduled visits, treatment plan, laboratory tests, and other study procedures.

Exclusion Criteria:

* Unresolved toxicity of Grade >1 attributed to prior therapies (excluding: Grade ≤2 neuropathy, alopecia, or skin pigmentation)
* Prior therapy with a WEE1 inhibitor
* A serious illness or medical condition(s).
* Pregnant or lactating females. Females of childbearing potential with a positive serum pregnancy test <14 days to Day 1.
* Subjects with active (uncontrolled, metastatic) second malignancies or requiring therapy.
* 12-lead ECG demonstrating a corrected QT interval using Fridericia's formula (QTcF) of >470 ms, except for subjects with atrioventricular pacemakers or other conditions (e.g., right bundle branch block) that render the QT measurement invalid.
* History or current evidence of congenital or family history of long QT syndrome or Torsades de Pointes (TdP).
* Taking medications with a known risk of TdP.
* Administration of strong and moderate CYP3A4 inhibitors/inducers and strong and moderate P-gp inhibitors.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 84 (Estimated)
Dates: Start 2021-08-01 (Actual); Primary Completion 2023-08-30 (Actual); Study Completion 2023-12-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of dose-limiting toxicities (DLT) in DLT evaluable subjects and the incidence and severity of adverse events. | Through Cycle 1 (21 days) Phase 1
Event-free survival (EFS) at 18 weeks per RECIST (Response Evaluation Criteria in Solid Tumors) Guideline version 1.1. | During phase 2, at 18 weeks
  EFS at 18 weeks is defined as time from study enrollment until date of disease progression, or detection of disease at a previously uninvolved site, or date of death of the subjects at 18 weeks.

SECONDARY OUTCOMES:
Event-free survival (EFS) per RECIST Guideline version 1.1. | At 12 months
  EFS is defined as time from study enrollment until date of last contact, date of disease progression, or detection of disease at a previously uninvolved site, or date of death.
Median overall survival (OS) and OS at 12 months per RECIST Guideline version 1.1. | At 12 months
  OS is defined as the time from date of first dosing until the date of death.
The frequency and severity of adverse events (AEs) and laboratory abnormalities per the National Cancer Institute Common Terminology (NCI CTCAE) version 5.0.lities. | Through completion, approximately 42 months
Plasma pharmacokinetics (PK) maximum concentration (Cmax). | Through completion, approximately 42 months
Plasma PK time to maximum concentration (Tmax). | Through completion, approximately 42 months
Area under the plasma concentration versus timepoint curve (AUC last). | Through completion, approximately 42 months
Terminal half-life of the plasma PK concentration. | Through completion, approximately 42 months

CONTACTS AND LOCATIONS:
Locations (17):
- United States (12):
  - Site 0106, Los Angeles, California
  - Site 0124, Oakland, California
  - Site 0195, Santa Monica, California
  - University of Florida College of Medicine, Gainesville, Florida
  - Site 0105, New York, New York
  - Site 0107, Cincinnati, Ohio
  - Site 0123, Portland, Oregon
  - Site 0193, Memphis, Tennessee
  - Site 0197, Nashville, Tennessee
  - Site 0103, Houston, Texas
  - Site 0188, Richmond, Virginia
  - Site 0122, Seattle, Washington
- France (5):
  - Site 3604, Bordeaux
  - Site 3601, Lyon
  - Site 3602, Marseille
  - Site 3606, Paris
  - Site 3605, Toulouse